CLINICAL TRIAL: NCT01774552
Title: A Pilot Study of Photo Acoustic Microscopy and Optical Coherence Tomography Imaging Technologies to Evaluate the Port-wine Stain Birthmark Treatment Before and After Pulsed Dye Laser Treatment.
Brief Title: Evaluate the Port-wine Stain Birthmark Treatment Before and After Pulsed Dye Laser Treatment
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Wangcun Jia, PhD., Research Scientist, University of California, Irvine
Other Study IDs: 20129094
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Port-wine Stain
MeSH Terms: conditions — Port-Wine Stain | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Port-wine stain: Photo Acoustic Microscopy and Optical Coherence tomography
  Interventions: Device: Photo Acoustic Microscopy and Optical Coherence tomography

INTERVENTIONS:
Device: Photo Acoustic Microscopy and Optical Coherence tomography — Photo Acoustic Microscopy and Optical Coherence tomography

SUMMARY:
Port-wine stain is a congenital, progressive vascular malformation of human skin involving post-capillary venules that occurs in an estimated 0.3% of children and can alter personality development and psychological in children.

DETAILED DESCRIPTION:
The researchers at University of California, Irvine and Washington University in Saint Louis are collaborating in this project and developes new multiple imaging devices call photoacoustic microscopy and optical coherence tomography imaging technologies can be use to evaluate the response of port-wine stain from Pulse Dye Laser treatment.

ELIGIBILITY:
Inclusion Criteria:

* All age with diagnosis of Port-wine stain

Exclusion Criteria:

* No diagnosis of Port-wine stain

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population will be selected from Beckman Laser Medical Clinic, UCI
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2012-12; Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
evaluate the port-wine stain birthmark | up to 12 months
  pulsed dye laser treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wancun Jia, PhD, Principal Investigator — Beckman Laser Institute, UCI
Locations (1):
- Beckman Laser Institute Medical Clinic, Irvine, California, United States